CLINICAL TRIAL: NCT04388605
Title: Assessing the Safety of Pregnancy In the CoRonavirus pandEmic: a Nationwide Prospective Study
Brief Title: Assessing the Safety of Pregnancy In the CoRonavirus (COVID-19) pandEmic
Acronym: ASPIRE
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 20-30559
Record Dates: First submitted 2020-05-07; First posted 2020-05-14 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Corona Virus Infection; COVID; Pregnancy Related; Early Pregnancy
Keywords: COVID-19; Pregnancy; Coronavirus
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Months
Biospecimen Retention: Samples Without DNA — At-home blood spot kits will be used for serology surveillance. Tests will occur weekly during the first trimester and monthly during the second and third trimesters of pregnancy. Covid-19 antibody serology and cytokine testing will be assayed using these blood spot cars.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective nationwide cohort study of pregnant women enrolled early in gestation and followed for Covid-19 exposure and infection, with follow up of obstetrical outcomes and infant development through the first year of life.

DETAILED DESCRIPTION:
ASPIRE is focused on the first trimester, a critical and vulnerable period when all of a baby's organ systems form and the placenta - the crucial connection between mom and baby - develops.

Currently, there are no data about the effects of COVID-19 infections in the first trimester. The study will provide critical information to:

1. Guide the care of pregnant women
2. Protect the safety of their babies and families
3. Help those considering pregnancy in the future understand what it means to be pregnant in this new era

The investigators are recruiting 10,000 women from the start of pregnancy and will track COVID-19 exposures using frequent serology testing. The investigators will collect information during and after the pregnancy to try to determine the effects of COVID 19 for mom and baby.

Participants will be asked to do the following throughout pregnancy:

* Submit frequent, quick (<1 minute each) symptom tracking reports using your mobile phone and/or computer.
* Collect finger-stick blood samples from home at several points throughout your pregnancy.
* Give permission to review medical records related to your pregnancy, delivery and baby's development.
* Complete questionnaires online about your health during your pregnancy and after delivery of your baby.

ELIGIBILITY:
Inclusion Criteria:

* Over age 18
* Participant is 4-10 weeks pregnant (gestation)

Exclusion Criteria:

- Male (biologically unable to achieve pregnancy)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators are recruiting 10,000 women from the start of pregnancy (4-10 weeks gestation) and will track COVID-19 exposures using frequent serology testing. The investigators will collect information during and after the pregnancy to try to determine the effects of COVID 19 for mom and baby.
Sampling Method: Non-Probability Sample
Enrollment: 7965 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of SARS-CoV-2 infection throughout pregnancy in women | Up to 9 months
  Determine the prevalence of SARS-CoV-2 infection throughout pregnancy in women whose pregnancy was documented at a SART member clinic in the United States between November 2019-December 2020. The investigators will use patient-reported information on infection symptoms as well as serological testing to capture both symptomatic and asymptomatic infections. Deliverable: By instituting the first prospectively tracked U.S.-based pregnancy cohort with precisely timed conception, the investigators will provide foundational, urgent data regarding the epidemiology of SARS-CoV-2 infection at varying gestational ages, across the real-time evolution of the COVID-19 pandemic and in the setting of various public health measures to reduce infection spread.
Incidence of SARS-CoV-2 infection throughout pregnancy in women | Up to 9 months
  Determine the incidence of SARS-CoV-2 infection throughout pregnancy in women whose pregnancy was documented at a SART member clinic in the United States between November 2019-December 2020. The investigators will use patient-reported information on infection symptoms as well as serological testing to capture both symptomatic and asymptomatic infections. Deliverable: By instituting the first prospectively tracked U.S.-based pregnancy cohort with precisely timed conception, the investigators will provide foundational, urgent data regarding the epidemiology of SARS-CoV-2 infection at varying gestational ages, across the real-time evolution of the COVID-19 pandemic and in the setting of various public health measures to reduce infection spread.

SECONDARY OUTCOMES:
Risk ratios of adverse obstetric in women infect with SARS-CoV-2 during early pregnancy onward compared to non-infected pregnant women | Up to 9 months
  Determine risk ratios of adverse obstetric outcomes in women infected with SARS-CoV-2 during early pregnancy onward compared to non-infected pregnant women. The investigators will focus on timing of infection (gestational month) and extent of COVID-19 symptoms as potential predictors of risk. Deliverable: The investigators will provide critical information about the maternal and fetal implications of SARS-CoV-2 infection at specific time points in pregnancy, compared to non-exposed pregnancies, and enable evidence-based obstetric surveillance protocols.
Risk ratios of adverse neonatal outcomes in women infected with SARS-CoV-2 during early pregnancy onward compared to non-infected pregnant women | Up to 1.5 years
  Determine risk ratios of adverse neonatal outcomes in women infected with SARS-CoV-2 during early pregnancy onward compared to non-infected pregnant women. The investigators will focus on timing of infection (gestational month) and extent of COVID-19 symptoms as potential predictors of risk. Deliverable: The investigators will provide critical information about the maternal and fetal implications of SARS-CoV-2 infection at specific time points in pregnancy, compared to non-exposed pregnancies, and enable evidence-based obstetric surveillance protocols.
Clinical, behavioral, and sociodemographic determinants | Up to 27 months
  Identify clinical, behavioral and sociodemographic determinants that predict risk of (a) maternal infection during pregnancy and (b) severe infection symptomatology (hospitalization, ICU admission). Deliverable: The investigators will provide novel findings that identify high-risk groups warranting more aggressive social avoidance measures during pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Huddleston, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Huddleston HG, Jaswa EG, Lindquist KJ, Kaing A, Morris JR, Hariton E, Corley J, Hoskin E, Gaw SL, Cedars MI. COVID-19 vaccination patterns and attitudes among American pregnant individuals. Am J Obstet Gynecol MFM. 2022 Jan;4(1):100507. doi: 10.1016/j.ajogmf.2021.100507. Epub 2021 Oct 11. No abstract available. PMID 34649015